CLINICAL TRIAL: NCT05045001
Title: Observational Retrospective Studies on Single Nucleotide Variants (SNPs) on the Interleukin-6 Receptor (IL6R) and Their Influence on the Response to Treatment and Safety in Patients With Specific Rheumatic Diseases
Brief Title: Pharmacogenetic Studies on Anti-IL-6 Receptor Monoclonal Antibodies on the Treatment of Rheumatic Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-IIL-2020-148
Record Dates: First submitted 2021-06-02; First posted 2021-09-16 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Rheumatoid Arthritis; Idiopathic Juvenile Arthritis; Giant Cell Arteritis; Still Disease
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Juvenile; Giant Cell Arteritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — DNA samples will be collected and stored following the appropriate national laws of Spain ( Ley de Investigación Biomédica 14/2007) regarding the use of human biological samples in biomedical investigation. Collection and storage approved by the organization's ethic committee.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Tocilizumab and Sarilumab are first-line biological disease-modifying anti-rheumatic drug (bDMARD) which inhibits Interleukin 6 (IL-6) pathway through blockade of its receptor on the treatment of Rheumatoid Arthritis and other rheumatic diseases as Giant Cell Arteritis, Still's disease and Idiopathic Juvenile Arthritis. At present, there is a lack of evidence to recommend the treatment of one bDMARD over another. Seeking for genetic biomarkers to predict response to treatment could be key towards a personalized treatment strategy in rheumatology.

The investigators aime to evaluate whether functional single nucleotide polymorphisms (SNPs) in the IL6R gene could predict response and/or toxicity in patients with rheumatic diseases treated with anti-IL-6 receptor drugs.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Rheumatoid Arthritis by the American College of Rheumatology (ACR) 2010 criteria or
* Diagnosis of Giant Cell Arteritis by the International League of Associations for Rheumatology (ILAR) criteria or
* Diagnosis of Still disease by classification criteria (Yamaguchi et al.) or
* Diagnosis of Idiopathic Juvenile Arthritis by ACR 1990 criteria.
* All of the previous must have been treated with anti-IL-6R monoclonal antibodies in the last 5 years

Exclusion Criteria:

* <18 years at recruitment
* Another rheumatic disease different of the ones in the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients being followed-up in the Hospital de la Santa Creu i Sant Pau, diagnosed of Rheumatoid Arthritis, Idiopathic Juvenile Arthritis, Still disease or Giant Cell Arteritis treated with anti-IL6R drugs.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2021-06-02 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
DAS28-C-reactive Protein (CRP) change | at 6 months
  Activity measure for patients with Rheumatoid Arthritis (RA)
Rate of adverse events | During treatment with anti-IL6R drugs
  Known adverse events during treatment with anti-IL6R drugs
CRP change | 6 months
  Acute phase reactant reduction in the other diseases different of RA.
Erythrocyte sedimentation rate (ESR) change | 6 months
  Acute phase reactant reduction in the other diseases different of RA.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Moya, Doctor, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No